CLINICAL TRIAL: NCT00797082
Title: Magnetic Resonance Diabetic Cardiac Stress Imaging : MRDIABETICS
Brief Title: Magnetic Resonance Diabetic Cardiac Stress Imaging
Acronym: MRDiabetics
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: default of inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: P070149; AOR07022 (Other: French Ministry)
Record Dates: First submitted 2008-10-27; First posted 2008-11-25 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Coronary Insufficiency
Keywords: Diabetic; Coronary disease; Atherosclerosis; Magnetic resonance imaging; Myocardial Perfusion Scintigraphy; Coronary angiography
MeSH Terms: conditions — Coronary Disease; Atherosclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): MRI = Myocardial Perfusion Stress and MPS = Myocardial Perfusion Scintigraphy
  * Diabetic patients
  * Coronary insufficiency
  Interventions: Device: MRI; Device: MPS

INTERVENTIONS:
Device: MRI — MRI = Myocardial Perfusion Stress
Device: MPS — MPS = Myocardial Perfusion Scintigraphy

SUMMARY:
The aim of the study is to assess the efficacy of cardiac MRI to detect coronary disease in diabetic patients. Cardiac MRI will be compared to myocardial scintigraphy with is the method being used in current practice. The investigators believe that cardiac MRI will be as efficient if not better that myocardial scintigraphy to detect tight coronary artery stenosis with the advantage of providing no radiation to the patient. Moreover, the investigators believe that cardiac MR will add additional information regarding possible undetected myocardial infarction.

DETAILED DESCRIPTION:
Rationale:

The incidence of diabetes is rising constantly. According to the WHO projections, the population of diabetics will double by 2025. In France, the current population of diabetics is estimated at 2.5 millions persons. The cause of death in diabetics involves a cardiovascular condition in approximately 65-80% of the cases. The leading event is myocardial infarction. The prevalence of silent myocardial ischemia (SMI) in diabetics varies widely from 10 to 30%. The prognosis of SMI is closely dependent on the presence or not of angiographically significant coronary artery stenosis - CAS (patients with SMI and CAS>70% show 31% of major cardiac events at 41±24 months vs only 1.4% in patients with SMI and no CAS>70%). It seems therefore important to identify diabetic patients with SMI and CAS especially knowing that endovascular or surgical treatments are available and can potentially improve the prognosis of such patients.

Myocardial Perfusion Scintigraphy (MPS) is widely prescribed to detect coronary stenosis. It has a high sensitivity (90%) but an intermediate specificity (75%), providing a significant amount of false positive cases. Such false positive cases are usually followed with unnecessary coronary angiographies. Myocardial Perfusion Stress MRI (MRI) has been recently developed and shows promising preliminary results (equivalent sensitivity, higher specificity compared to MPS) for the identification of coronary artery stenosis. Few studies directly compare MRI and MPS in the general population, none in the diabetic population.

Principal objective: To evaluate and compare diagnostic performances of MRI and MPS for the diagnosis of coronary insufficiency in diabetic patients free of known coronary disease.

Secondary objective:

* Cost efficacy analysis for the diagnosis of coronary insufficiency in diabetic patients free of known coronary disease.
* Impact of clinical information on MRI and MPS diagnostic performances.

Design:. Prospective, monocentric study, where MRI and MPS will be assessed in a centralised manner by 2 independent blinded readers (2 readers for each technique) and compared to coronary angiography (Gold Standard, assessed by 2 independent blinded readers).

Patient selection: Patient with diabetes (type 1 or type 2), free of known coronary disease, addressed for MPS.

Inclusion period length: 24 months

Follow up period length: 2 days

Principal judgement criteria:

Coronary angiography: positive diagnosis of CAS if stenosis >50% on the left coronary artery (trunk) or stenosis >70% on the IVA (inter ventricular artery), LCx (circumflex artery) or RCA (right coronary artery) and branches.

MPS : positive diagnosis of CAS based on the following criteria : severity perfusion index, reversibility, contractility anomalies, signal attenuation due to patient morphology.

MRI : positive diagnosis of CAS based on an algorithm including the following criteria : first pass perfusion defect at stress, reversibility at rest, Myocardial Delayed Enhancement.

Number of necessary patients: 165

Expected results: An assessment of MRI performances compared to MPS for the diagnosis of coronary insufficiency in diabetic patients free of known coronary disease that will help improve diagnostic strategy.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patient older than 18 years old
* Patient with health care coverage ( social security or universal health coverage - CMU)
* Patient who had a prior medical examination
* Diabetic patient (type 1 or type 2) with no known coronary artery disease, addressed for myocardial scintigraphy
* Patient who was informed of objectives and constraints of the study and having given his consent in writing

EXCLUSION CRITERIA:

* Pregnant and lactating women
* Patients with known coronary disease (myocardial infarction, unstable angina, history of coronary artery disease)
* Patient with contra-indication for MRI claustrophobia, metallic foreign body in the eye, pacemakers, mechanical heart valve laid before 1985 Patient with specific contra-indication to vasodilators
* Severe hypotension < 90 mmHg
* Hypersensitivity to adenosine or dipyridamole
* Bronchial asthma, chronic obstructive pulmonary disease with obvious bronchospasm. Severe and known pulmonary artery hypertension
* Atrioventricular 2nd or 3rd degree blocks, long QT syndrome
* Tight known carotid artery stenosis (70% NASCET criterion), with no possible vascular substitution
* Patient with contra-indication to cardiac stimulation
* Unstable hemodynamic state and / or unstable angina not stabilized by drug treatment and/or decompensated or severe heart failure
* Known comorbidities : pregnancy and lactation, tight aortic valve or mitral valve stenosis, severe left-right shunt, severe pericarditis or abundant pericardial effusion
* Contra-indication to coronary angiography
* Renal failure with creatinine clearance < 30 ml / min
* Hypersensitivity to contrast agents that resulted in a serious complication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-11; Primary Completion 2011-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
positive diagnosis of coronary artery disease. | 2 days

SECONDARY OUTCOMES:
cost efficacy analysis for the diagnosis of coronary insufficiency in diabetic patients free of known coronary disease | 26 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Michel SERFATY, PHU, Principal Investigator — ASSISTANCE PUBLIQUE
Locations (1):
- Hopital Bichat, Paris, France